CLINICAL TRIAL: NCT02696564
Title: Losartan Effects on Emphysema Progression
Acronym: LEEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U01HL128951 (NIH)
Record Dates: First submitted 2016-02-25; First posted 2016-03-02 (Estimated); Results first posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Emphysema
Keywords: COPD; emphysema; HRCT; losartan
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Losartan (Active Comparator): At randomization participants will start with a dose of 50mg (one capsule) once a day for 2 weeks. If this dose is well tolerated and systolic BP is >90 mm Hg and diastolic BP is > 60 mm Hg, the dose will be increased to 100 mg (2 capsules) once a day for the remaining 46 weeks.
  Interventions: Drug: Losartan
- placebo (Placebo Comparator): At randomization participants will start with a dose of one capsule (inactive) once a day for 2 weeks. After two weeks, if systolic BP is >90 mm Hg and diastolic BP is > 60 mm Hg, the dose will be increased to 2 capsules once a day for the remaining 46 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — 50mg once per day for two weeks,followed by 100mg once per day for 46 weeks if increased dose tolerated
  Arms: Losartan
Drug: Placebo — one capsule per day for two weeks, followed by two capsules per day for 46 weeks
  Arms: placebo

SUMMARY:
A randomized, parallel, placebo controlled trial to evaluate the effect of 100mg/day losartan on the progression of emphysema as measured by quantitative HRCT compared to placebo

.

DETAILED DESCRIPTION:
This is a trial designed to test if a treatment, losartan, may decrease the progression of Chronic Obstructive Pulmonary Disease (COPD). Losartan is an angiotensin receptor blocking agent, commonly used as an antihypertensive agent, which has been shown to alter cardiac remodeling after myocardial infarction and renovascular remodeling in diabetes-mellitus. In this trial participants with mild to severe COPD, with Computed Tomography (CT) evidence of emphysema (5-35% of voxels with < -950 Hounsfield Units), will be randomly assigned to receive 100mg/day of losartan or placebo for 48 weeks. The primary outcome measure will be the rate of progression of emphysema, quantified as the percent of lung voxels with a density less than -950 HU as measured by High Resolution CT (HRCT, from baseline to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Mild to severe COPD: Ratio of forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) less than or equal to 0.70, FEV1 20-80% of predicted
* Current or former smoker
* HRCT scan with 5-35% of voxels with density less than -950 Hounsfield Units (HU)
* Ability to understand and willingness to sign consent documents

Exclusion Criteria:

* Current therapy with angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB)
* Known intolerance to ACE inhibitor or ARB
* History of angioedema
* Conventional indication for ACE inhibitor or ARB (e.g., history of myocardial infarction, known cardiomyopathy)
* Renal insufficiency (GFR <30 mL/min by Cockcroft-Gault calculation)
* Current regular use of NSAIDs defined as daily use 5 or more days of the week for more than one month
* Potassium supplementation or serum potassium level of 5.0 milliequivalents (mEq)/dL or higher at V1
* Current use of a potassium sparing diuretic
* COPD exacerbation requiring treatment within 6 weeks at V1
* Chronic systemic corticosteroid use of more than 10mg/day of prednisone
* Resting SpO2 <89% on 2 L nasal cannula continuous flow; unless at altitude > 4,000 feet, then resting oxygen saturation (SpO2) <89% on 4 L N C continuous flow
* Untreated arterial hypertension (systolic blood pressure greater than140 mm Hg, diastolic blood pressure greater than 90 mm Hg)
* Blood pressure less than 90 mm Hg systolic or 60 mm Hg diastolic while standing or sitting
* Known unilateral or bilateral renal artery stenosis higher than 70%
* Previous lung resection surgery
* Evidence of interstitial, occupational or chronic infectious lung disease
* Changes to chest that preclude adequate HRCT imaging (e.g. Metallic objects in the chest such as shrapnel or pacemaker leads)
* For women of child bearing potential, positive pregnancy test or unwillingness to use two methods of birth control or abstinence for the duration of the study
* Major chronic illnesses which in the judgment of the study physician would interfere with participation in the study e.g. including but not limited to: cardiac, renal, hepatic (LFTs more than 2.5x normal upper limit), neurological, psychiatric, endocrine or neoplastic diseases, uncontrolled diabetes, uncontrolled HIV infection or other immune system disorder, hyperthyroidism, seizure disorders, non-skin cancer, rheumatic diseases
* Failure to keep screening appointments or other indicators of non-adherence
* Inability to be contacted by telephone
* Intention to leave area within 12 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wise, MD, Principal Investigator — Johns Hopkins University; Janet Holbrook, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of California at San Diego, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Western Connecticut Health Network, Danbury, Connecticut
  - University of Florida College of Medicine, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Hospitals, Chicago, Illinois
  - St. Vincent Hospital and Health Care Center, Inc., Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Louisiana State University, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - St. Louis University School of Medicine, St Louis, Missouri
  - St. Louis Asthma Clinical Research Center - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai National Jewish Health Respiratory Institute; Icahn School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Vermont Lung Center at The University of Vermont, Colchester, Vermont
  - Pacific Northwest Airways - VA Puget Sound Healthcare System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC)

REFERENCES:
- [Derived] Wise RA, Holbrook JT, Brown RH, Criner GJ, Dransfield MT, He J, Henderson RJ, Kaminsky DA, Kaner RJ, Lazarus SC, Make BJ, McCormack MC, Neptune ER, Que LG. Clinical Trial of Losartan for Pulmonary Emphysema: Pulmonary Trials Cooperative Losartan Effects on Emphysema Progression Clinical Trial. Am J Respir Crit Care Med. 2022 Oct 1;206(7):838-845. doi: 10.1164/rccm.202201-0206OC. PMID 35649189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2,779 individuals were screened for this study; of those, 2,028 were determined to be ineligible, and 531 declined to participate.
Pre-assignment Details: 220 individuals were randomized into the study.
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 108 | 112
Completed | 94 | 99
Not Completed | 14 | 13
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Missed final HRCT scan due to coronavirus disease pandemic | 3 | 1
Not completed — Baseline and final high-resolution computed tomography (HRCT) scans conducted on different scanners | 2 | 2
Not completed — High-resolution computed tomography (HRCT) scan conducted on unknown scanner | 1 | 1
Not completed — Participant diagnosed with lung cancer | 1 | 0
Not completed — Incorrect kernel used in high-resolution computed tomography (HRCT) scan | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 108 | 112 | 220
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [63 to 74] | 65 [61 to 71] | 65 [61 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 93
  Male | 61 | 66 | 127
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 19 | 23 | 42
  White | 88 | 88 | 176
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 108 | 112 | 220
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 27 [22 to 31] | 26 [23 to 28] | 26 [23 to 29]
Current smokers (past month) [Count of Participants; unit: Participants] | 26 | 26 | 52
Smoking history [Median (Inter-Quartile Range); unit: Pack-years] | 46 [35 to 60] | 42 [34 to 57] | 44 [34 to 58]
Spirometry percent predicted [Median (Inter-Quartile Range); unit: Percent predicted] — Population: Pre-bronchodilator spirometry results were not available for 11 participants in the Losartan group and 8 participants in the Placebo group.
  Percent predicted
    Pre-bronchodilator % predicted FEV1: number analyzed (Participants) | 97 | 104 | 201
    Pre-bronchodilator % predicted FEV1 | 43 [33 to 57] | 43 [31 to 54] | 43 [33 to 55]
    Post-bronchodilator % predicted FEV1 | 48 [37 to 61] | 48 [35 to 59] | 48 [36 to 59]
Spirometry pre-bronchodilator FEV1 [Median (Inter-Quartile Range); unit: Liters] — Population: Pre-bronchodilator spirometry results were not available for 11 individuals from the Losartan group and 8 individuals from the Placebo group.
  Liters
    number analyzed (Participants) | 97 | 104 | 201
    (all) | 1.1 [0.9 to 1.5] | 1.1 [0.8 to 1.5] | 1.1 [0.9 to 1.5]
Sitting Blood Pressure [Median (Inter-Quartile Range); unit: Millimeters of mercury (mmHg)]
  Systolic | 125 [116 to 133] | 123 [111 to 134] | 124 [113 to 133]
  Diastolic | 77 [72 to 81] | 75 [68 to 81] | 76 [70 to 81]
St. George's Respiratory Questionnaire for chronic obstructive pulmonary disease (COPD) score [Median (Inter-Quartile Range); unit: units on a scale] — The St George's Respiratory Questionnaire for COPD patients (SGRQ-C) is a 40-item questionnaire designed to measure impact on overall health, daily life, and perceived well-being in patients with COPD. The SGRQ-C includes three categories: Symptoms (frequency and severity), Activities caused or limited by breathlessness, and Impacts on social and psychological functioning caused by airways disease. The total score and scores for each category range from 0 to 100, with higher scores indicating more limitations.
  units on a scale
    Total | 42 [30 to 52] | 40 [26 to 61] | 42 [28 to 55]
    Symptoms | 55 [39 to 71] | 56 [37 to 73] | 55 [39 to 72]
    Activity | 59 [46 to 66] | 59 [43 to 79] | 59 [46 to 72]
    Impact | 28 [14 to 41] | 26 [14 to 45] | 27 [14 to 42]
COPD Assessment Test [Median (Inter-Quartile Range); unit: units on a scale] — The COPD Assessment Test (CAT) is an 8-item questionnaire assessing the impact of COPD on health status. CAT scores range from 0 to 40, with higher scores indicating a more severe impact of COPD on a patient's life. Scores of 0 to 10 are classified as "Mild", scores of 11 to 20 are classified as "Moderate", 21 to 30 indicates a "Severe" score, and 31 to 40 is a "Very Severe" score.
  units on a scale | 17 [13 to 22] | 16 [11 to 25] | 17 [12 to 23]
COPD Assessment Test impact level [Count of Participants; unit: Participants] — The COPD Assessment Test (CAT) is an 8-item questionnaire assessing the impact of COPD on health status. CAT scores range from 0 to 40, with higher scores indicating a more severe impact of COPD on a patient's life. Scores of 0 to 10 are classified as "Mild", scores of 11 to 20 are classified as "Moderate", 21 to 30 indicates a "Severe" score, and 31 to 40 is a "Very Severe" score.
  Participants
    Mild | 21 | 26 | 47
    Moderate | 52 | 45 | 97
    Severe | 35 | 33 | 68
    Very severe | 0 | 8 | 8
Modified Medical Research Council dyspnea scale [Median (Inter-Quartile Range); unit: units on a scale] — The modified Medical Research Council dyspnea scale (mMRC) is a self-rating tool to measure how much breathlessness affects someone's day to day activities. Scores are between 0 and 4, with higher scores indicating more severe breathlessness.
  units on a scale | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
PROMIS Physical Function-20a [Median (Inter-Quartile Range); unit: units on a scale] — The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 20a is a 20-item questionnaire used to indicate a patient's ability to perform activities of daily living, such as bathing, dressing, and commuting. Raw scores from this questionnaire are compared to a reference population to create a "T-score". The general US population is the reference population. In this T-score metric, 50 indicates the population mean with a standard deviation or 10. Higher scores mean better outcomes (more ability to do activities of daily living).
  units on a scale | 40 [38 to 44] | 40 [36 to 44] | 40 [37 to 44]

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean pct950
Description: change in percentage of voxels with density less than -950 Hounsfield Units
Time Frame: 48 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of voxels
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 94 | 99
percentage of voxels | 1.35 [0.67 to 2.02] | 0.66 [0.09 to 1.23]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — We will estimate a 95% confidence interval for the losartan vs placebo mean difference, using the regression estimate and the t-distribution; we will reject the null that losartan is equivalent to placebo if the 95% interval excludes 0.0; p = 0.133, Mixed Models Analysis; P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

2. Secondary Outcome: Change From Baseline in Pre-bronchodilator FEV1 Percent Predicted
Description: Change from the first visit to the final visit in a spirometry (breathing test) measure: forced expiratory volume in one second (FEV1). The test is administered without the participant taking any bronchodilator medication. The FEV1 is compared to standard predicted values in the US population for each individual based on their height, gender, and ethnic group; the result is given as percent of predicted value.
Time Frame: 48 weeks
Population: Pre-bronchodilator results were not available at the baseline and/or final visit for 57 participants in the Losartan group and 56 participants in the placebo group. This was due in part to the elimination of all non-medically necessary spirometry testing during the COVID-19 pandemic.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of predicted value
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 51 | 56
percentage of predicted value | -0.99 [-3.18 to 1.20] | -0.54 [-2.47 to 1.38]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.762, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

3. Secondary Outcome: Change From Baseline in Post-bronchodilator FEV1 Percent Predicted
Description: Change from the first visit to the final visit in a spirometry (breathing test) measure: forced expiratory volume in one second (FEV1). This test is performed after the participant is given bronchodilator medications. The FEV1 is compared to standard predicted values in the US population for each individual based on their height, gender, and ethnic group; the result is given as percent of predicted value.
Time Frame: 48 weeks
Population: Post-bronchodilator results were not available at the baseline and/or final visit for 35 participants in the Losartan group and 39 participants in the placebo group. This was due in part to the elimination of all non-medically necessary spirometry testing during the COVID-19 pandemic.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of predicted value
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 73 | 73
percentage of predicted value | -2.60 [-4.22 to -0.98] | -2.37 [-3.71 to -1.03]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.834, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

4. Secondary Outcome: Change From Baseline in CAT Score
Description: Change from the first visit to the final visit in the participant's COPD Assessment Test (CAT) score. The CAT is an 8-item questionnaire assessing the impact of COPD on health status. CAT scores range from 0 to 40, with higher scores indicating a more severe impact of COPD on a patient's life.
Time Frame: 48 weeks
Population: CAT results were not available at the baseline and/or final visit for 9 participants in the Losartan group and 8 participants in the placebo group.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 99 | 104
score on a scale | -0.18 [-1.21 to 0.85] | 0.03 [-1.04 to 1.09]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.783, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

5. Secondary Outcome: Change From Baseline in SGRQ Score: Total
Description: Change from the first visit to the final visit in participants' score on the St George's Respiratory Questionnaire - COPD. The St George's Respiratory Questionnaire for COPD patients (SGRQ-C) is a 40-item questionnaire designed to measure impact on overall health, daily life, and perceived well-being in patients with COPD. The SGRQ-C includes three categories: Symptoms (frequency and severity), Activities caused or limited by breathlessness, and Impacts on social and psychological functioning caused by airways disease. The total score and scores for each category range from 0 to 100, with higher scores indicating more limitations.
Time Frame: 48 weeks
Population: Total SGRQ results were not available at the baseline and/or final visit for 9 participants in the Losartan group and 9 participants in the placebo group.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 99 | 103
score on a scale | -1.31 [-3.15 to 0.52] | 1.20 [-0.68 to 3.08]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.053, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

6. Secondary Outcome: Change From Baseline in SGRQ Score: Symptoms
Description: Change from the first visit to the final visit in participants' scores on the symptom-related questions on the St Georges Respiratory Questionnaire-COPD. The St George's Respiratory Questionnaire for COPD patients (SGRQ-C) is a 40-item questionnaire designed to measure impact on overall health, daily life, and perceived well-being in patients with COPD. The SGRQ-C includes three categories: Symptoms (frequency and severity), Activities caused or limited by breathlessness, and Impacts on social and psychological functioning caused by airways disease. The total score and scores for each category range from 0 to 100, with higher scores indicating more limitations.
Time Frame: 48 weeks
Population: SGRQ results were not available at the baseline and/or final visit for 9 participants in the Losartan group and 9 participants in the placebo group.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 99 | 103
score on a scale | -6.19 [-8.76 to -3.62] | -1.78 [-4.04 to 0.49]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.016, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

7. Secondary Outcome: Change From Baseline in SGRQ Score: Activity
Description: Change from the first visit to the final visit in participants' scores on the activity-related questions on the St Georges Respiratory Questionnaire-COPD. The St George's Respiratory Questionnaire for COPD patients (SGRQ-C) is a 40-item questionnaire designed to measure impact on overall health, daily life, and perceived well-being in patients with COPD. The SGRQ-C includes three categories: Symptoms (frequency and severity), Activities caused or limited by breathlessness, and Impacts on social and psychological functioning caused by airways disease. The total score and scores for each category range from 0 to 100, with higher scores indicating more limitations.
Time Frame: 48 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 99 | 103
score on a scale | -0.66 [-3.22 to 1.91] | 2.45 [-0.10 to 5.00]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.065, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

8. Secondary Outcome: Change in SGRQ Score: Impact
Description: Change from the first visit to the final visit in participants' scores on the impact-related questions on the St Georges Respiratory Questionnaire-COPD. The St George's Respiratory Questionnaire for COPD patients (SGRQ-C) is a 40-item questionnaire designed to measure impact on overall health, daily life, and perceived well-being in patients with COPD. The SGRQ-C includes three categories: Symptoms (frequency and severity), Activities caused or limited by breathlessness, and Impacts on social and psychological functioning caused by airways disease. The total score and scores for each category range from 0 to 100, with higher scores indicating more limitations.
Time Frame: 48 weeks
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 99 | 103
score on a scale | -0.25 [-2.46 to 1.96] | 1.35 [-0.67 to 3.38]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.293, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

9. Secondary Outcome: Change From Baseline in mMRC Dyspnea Scale
Description: Change from the first visit to the final visit in participants' scores on the modified Medical Research Council dyspnea scale. The modified Medical Research Council dyspnea scale (mMRC) is a self-rating tool to measure how much breathlessness affects someone's day to day activities. Scores are between 0 and 4, with higher scores indicating more severe breathlessness.
Time Frame: 48 weeks
Population: mMRC dyspnea scale results were not available at the baseline and/or final visit for 9 participants in the Losartan group and 9 participants in the placebo group.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 99 | 103
score on a scale | 0.01 [-0.15 to 0.16] | 0.11 [-0.03 to 0.26]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.356, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

10. Secondary Outcome: Change From Baseline in PROMIS-20a T-score
Description: Change from the first visit to the final visit in participants' scores on the Patient-Reported Outcome Measures Information System (PROMIS) Physical Function assessment. The Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form 20a is a 20-item questionnaire used to indicate a patient's ability to perform activities of daily living, such as bathing, dressing, and commuting. Raw scores from this questionnaire are compared to a reference population to create a "T-score". The general US population is the reference population. In this T-score metric, 50 indicates the population mean with a standard deviation of 10. Higher scores mean better outcomes (more ability to do activities of daily living)
Time Frame: 48 weeks
Population: PROMIS-20a results were not available at the baseline and/or final visit for 9 participants in the Losartan group and 10 participants in the placebo group.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 99 | 102
score on a scale | 0.00 [-0.59 to 0.59] | -1.04 [-1.62 to -0.45]
Statistical Analysis 1: Comparison: Losartan vs Placebo; Test type: Superiority — Statistical differences were inferred if the 95% confidence intervals (CI) did not include zero; p = 0.009, Mixed Models Analysis — P-value based on generalized linear mixed models with covariates for site, baseline value, and for treatment group

11. Post Hoc Outcome: Number of COPD Exacerbations by Severity and Treatment Assignment
Description: This measure assessed the number of exacerbations of chronic obstructive pulmonary disease in both the losartan and placebo treatment groups. Participants were asked about current and past exacerbations during each study visit. Exacerbations were defined as 2 or more worsening COPD symptoms lasting 3 or more consecutive days that required a new prescribed treatment. Each exacerbation was further classified as "mild" (requiring only a change in existing COPD medications),"moderate" (requiring a new prescription for a steroid and/or antibiotic), or "severe" (requiring a hospitalization for COPD symptoms).
Time Frame: 48 weeks
Population: The analysis population consists of the number of participants who reported at least one exacerbation in each treatment group. Two participants in the losartan treatment group did not report any COPD exacerbations during the study.
Measure: Number; unit: exacerbation events
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 106 | 112
exacerbation events
  Mild exacerbation | 3 | 4
  Moderate exacerbation | 41 | 47
  Severe exacerbation | 7 | 21
Statistical Analysis 1: Comparison: Losartan vs Placebo; P-value for rate of mild exacerbations between treatment groups (measured in events per 100 person-years); Test type: Superiority; p = 0.892, Negative binomial model; Relative rate (losartan to placebo) = 0.80, 95% CI 2-sided [0.03 to 18.77]
Statistical Analysis 2: Comparison: Losartan vs Placebo; P-value for rate of moderate exacerbations between treatment groups (measured in events per 100 person-years); Test type: Superiority; p = 0.946, Negative binomial model; Relative rate (losartan to placebo) = 0.91, 95% CI 2-sided [0.05 to 14.97]
Statistical Analysis 3: Comparison: Losartan vs Placebo; P-value for rate of severe exacerbations between treatment groups (measured in events per 100 person-years); Test type: Superiority; p = 0.487, Negative binomial model; Relative rate (losartan to placebo) = 0.36, 95% CI 2-sided [0.02 to 6.51]

ADVERSE EVENTS:
Time Frame: Baseline up to 48 weeks
Description: Adverse events were assessed throughout the study through regular physical exams by a study physician, symptom questionnaires and medical history review at each study visit, and blood testing at the beginning, middle, and end of the study.
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 1/108 | 2/112
Serious Adverse Events (participants affected / at risk) | 18/108 | 25/112
Other Adverse Events (participants affected / at risk) | 106/108 | 112/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=108) | Placebo (N=112)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 15 (19)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Acute respiratory failure secondary to end stage COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Collapsed lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Radiation pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 3 (3)
Total knee replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal fusion revision (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Falls (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dehydration (General disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Near syncope (Nervous system disorders) | 0 (0) | 1 (1)
Pseudogout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=108) | Placebo (N=112)
Chest pain (Cardiac disorders) | 9 (10) | 8 (9)
Edema (Skin and subcutaneous tissue disorders) | 8 (9) | 10 (15)
Skin rash or hives (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (9)
Diarrhea (Gastrointestinal disorders) | 13 (15) | 12 (16)
Heartburn/indigestion (Gastrointestinal disorders) | 11 (17) | 24 (36)
Nausea/vomiting (Gastrointestinal disorders) | 7 (7) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (57) | 38 (77)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 28 (46) | 30 (49)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 30 (50) | 32 (63)
Weakness (Musculoskeletal and connective tissue disorders) | 19 (36) | 24 (36)
Dizziness/lightheadedness (Nervous system disorders) | 27 (34) | 16 (20)
Headache/ head pain (Nervous system disorders) | 26 (38) | 35 (52)
Fatigue (General disorders) | 38 (71) | 41 (77)
Fever (General disorders) | 5 (5) | 6 (6)
Sleep problems (General disorders) | 30 (46) | 34 (65)
Sore throat (General disorders) | 8 (9) | 18 (24)
Congestion (Respiratory, thoracic and mediastinal disorders) | 42 (73) | 47 (70)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 34 (57)
Mild COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Moderate COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 25 (41) | 29 (47)
Severe COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 14 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT02696564/Prot_SAP_000.pdf